CLINICAL TRIAL: NCT01355380
Title: The Efficacy of Inhaled Iloprost in Patients Treated Within the "Pulmonary Arterial Hypertension Therapeutic Programme".
Brief Title: Efficacy of Ventavis Used in Real-life Setting.
Acronym: SPHERA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15308; VE1010PL (Other: Company internal)
Record Dates: First submitted 2011-05-17; First posted 2011-05-18 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension; Inhaled iloprost; Quality of life
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Iloprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Drug (incl. Placebo)
  Interventions: Drug: Inhaled iloprost (Ventavis, BAYQ6256)

INTERVENTIONS:
Drug: Inhaled iloprost (Ventavis, BAYQ6256) — Patients treated with inhaled iloprost (Ventavis) 2.5 or 5 micrograms 6-9 times daily

SUMMARY:
This is a registry of patients diagnosed with pulmonary arterial hypertension, scheduled for treatment with Ventavis.

Typical clinical measures and quality of life will be prospectively followed in 12 months period.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary arterial hypertension in WHO functional class III or IV
* Age 18+
* Patients newly treated with Ventavis or switched from sildenafil

Exclusion Criteria:

* Retrospective documentation is not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients prescribed Ventavis within the Pulmonary Arterial Hypertension Therapeutic Programme.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2010-08-05 (Actual); Primary Completion 2016-04-28 (Actual); Study Completion 2016-09-22 (Actual)

PRIMARY OUTCOMES:
Changes of the exercise capacity as measured by 6-minutes walking distance | 3, 6, 9 and 12 months vs. baseline

SECONDARY OUTCOMES:
Changes of depression score over time | 3, 6, 9 and 12 months vs. baseline
Changes of functional capacity as measured by WHO classification system | 3, 6, 9 and 12 months vs. baseline
Changes of pulmonary haemodynamics | 3, 6, 9 and 12 months vs. baseline
Changes of serum level of natriuretic peptide B | 3, 6, 9 and 12 months vs. baseline
Changes of Quality of Life score | 3, 6, 9 and 12 months vs. baseline
Changes in cardiac echo parameters | 3, 6, 9 and 12 months vs. baseline
Number of patients with treatment-emergent adverse events | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Poland